CLINICAL TRIAL: NCT04017455
Title: Neoadjuvant Treatment in Rectal Cancer With Radiotherapy Followed by Atezolizumab and Bevacizumab (TARZAN)
Acronym: TARZAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N18TRZ
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer
Keywords: short term immunotherapy; atezolizumab; bevacizumab; radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: single group, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- bevacizumab and atezolizumab (Experimental): 1 cycle of bevacizumab monotherapy, followed by 2 cycles of bevacizumab combined with atezolizumab, followed by 1 cycle of atezolizumab monotherapy
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — 3 cycles of atezolizumab 840 mg
  Other Names: MPDL3280A
Drug: Bevacizumab — 3 cycles of bevacizumab 5mg/kg
  Other Names: HCA 185 ,Avastin

SUMMARY:
In this study, patients with resectable rectal cancer will receive radiotherapy, followed by neoadjuvant bevacizumab and atezolizumab

DETAILED DESCRIPTION:
38 patients with resectable rectal cancer will be enrolled. All patients will be treated with radiotherapy followed by bevacizumab and atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients age 18 years and older
* histologically confirmed adenocarcinoma of the rectum
* intermediate risk rectal cancer or low risk distal rectal cancer

Exclusion Criteria:

* evidence of metastatic disease
* prior radiation therapy for disease under study
* prior treatment with CD137 agonists or immune checkpoint blockade therapies
* current or recent use of acetylsalicylic acid
* history of clinically significant cardiac or pulmonary dysfunction pregnancy or breastfeeding
* significant auto-immune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
clinical complete and near-complete response rate | 12 weeks post-radiotherapy
  response rate will be assessed by MRI and endoscopy

SECONDARY OUTCOMES:
incidence of adverse events following treatment (safety) | untill 100 days after last patient last study drug
  adverse events will be assessed (according tot CTC-AE v5) during treatment
local recurrence rate at 1 year follow-up | 1 year post-radiotherapy
  recurrence will be assessed by MRI and CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Chalabi, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Marieke van de Belt, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No